CLINICAL TRIAL: NCT07395817
Title: Feasibility and Preliminary Effectiveness of Video Conference-Based Brief Cognitive Behavioral Therapy (V-BCBT) for Outpatients With Mood Disorders at High Risk for Suicide: A Pilot Randomized Controlled Trial
Brief Title: Video Conference-Based Brief Cognitive Behavioral Therapy for Suicidal High-Risk Outpatients With Mood Disorders
Acronym: V-BCBT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hyung Keun Park (Other)
Responsible Party: Sponsor-Investigator, Hyung Keun Park, Clinical Assistant Professor, Department of Psychiatry, Asan Medical Center
Organization: Asan Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2026-0177
Record Dates: First submitted 2026-02-01; First posted 2026-02-09 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Suicidal Ideation and Behaviors; Suicide Attempt; Cognitive Behavioral Therapy
Keywords: Suicidal Ideation and Behaviors; Suicide Attempt; Cognitive Behavioral Therapy for Suicidality
MeSH Terms: conditions — Suicidal Ideation; Behavior; Suicide, Attempted | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Videoconference-Based Brief Cognitive Behavioral Therapy (V-BCBT) + Treatment as Usual (TAU) (Experimental): Participants in this arm will receive Videoconference-Based Brief Cognitive Behavioral Therapy (V-BCBT) in addition to Treatment as Usual (TAU) provided in the outpatient setting. After randomization, they will complete 8 individual videoconference sessions of V-BCBT (approximately 50 minutes per session, twice weekly for 4 weeks), while continuing to receive routine outpatient care. TAU may include pharmacotherapy and supportive psychotherapy as typically provided in outpatient psychiatric services.
  Interventions: Behavioral: Videoconference-Based Brief Cognitive Behavioral Therapy (V-BCBT); Other: Treatment as Usual (TAU)
- Treatment as Usual (TAU) only (Active Comparator): Participants in this arm will receive Treatment as Usual (TAU) only through outpatient psychiatric services. TAU is delivered according to clinical need and may include pharmacotherapy and supportive psychotherapy as routinely provided.
  Interventions: Other: Treatment as Usual (TAU)

INTERVENTIONS:
Behavioral: Videoconference-Based Brief Cognitive Behavioral Therapy (V-BCBT) — Behavioral: V-BCBT is a brief, structured cognitive behavioral therapy (CBT) program delivered via videoconference for suicidal high-risk outpatients with mood disorders. It aims to reduce post-treatment and follow-up suicide risk by improving crisis coping/self-regulation, strengthening reasons for living, and shifting maladaptive "suicide mode" responses to adaptive alternatives. It includes 8 individual sessions (approximately 50 minutes) in three phases: (1) Crisis management (1-2): alliance, psychoeducation, crisis response plan (warning signs, coping, supports/resources), hope kit, and means safety; (2) Skills (3-6): relaxation, sleep regulation, behavioral activation/values goals, cognitive restructuring, mindfulness; (3) Relapse prevention (7-8): skills review, coping rehearsal, and a relapse prevention plan (update crisis plan). Sessions include practice and homework.
  Other: TAU is routine outpatient care as indicated (e.g., medication and supportive psychotherapy).
  Arms: Videoconference-Based Brief Cognitive Behavioral Therapy (V-BCBT) + Treatment as Usual (TAU)
Other: Treatment as Usual (TAU) — Treatment as Usual (TAU) refers to routine outpatient care provided as clinically indicated, including medication treatment and supportive psychotherapy.

SUMMARY:
This pilot randomized controlled trial aims to evaluate the feasibility, acceptability, and preliminary effectiveness of videoconference-based brief cognitive behavioral therapy (V-BCBT) for adult outpatients with mood disorders who are at high risk for suicide. Eligible participants will be randomized (1:1) to either V-BCBT + treatment as usual (TAU) or TAU alone. V-BCBT consists of eight structured videoconference sessions (approximately 50-60 minutes each, twice weekly for 4 weeks) focusing on crisis management (for example, understanding the "suicide mode," developing a crisis response plan, strengthening reasons for living), cognitive and behavioral coping skills (for example, relaxation, behavioral activation, cognitive restructuring, mindfulness), and relapse prevention (for example, coping rehearsal and a relapse prevention plan).

ELIGIBILITY:
Inclusion Criteria:

* High suicide risk, defined as either (a) a suicide attempt within the past 1 month or (b) Beck Scale for Suicide Ideation (SSI) ≥ 5.
* Aged 18 years or older.
* Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) diagnosis of a depressive disorder or bipolar and related disorder, confirmed at screening using the Mini International Neuropsychiatric Interview (M.I.N.I.).
* Able to read and write Korean without difficulty.
* Has access to a device (e.g., computer, tablet, or smartphone) and internet connectivity to participate in remote intervention.
* Able to understand the study, voluntarily provide written informed consent, and agree to comply with study procedures/precautions.

Exclusion Criteria:

* Currently in an activated manic state with psychotic symptoms, or has a severe psychiatric disorder (e.g., schizophrenia spectrum disorder), or a clinically significant neurological disorder, brain injury, intellectual disability, or any other medical condition that would prevent study participation.
* Has received psychotherapy within 3 months prior to screening (e.g., CBT, interpersonal psychotherapy, psychodynamic psychotherapy, or psychoanalysis).
* Is in an acute suicidal crisis requiring immediate inpatient hospitalization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Suicide Attempts from Baseline to 3 Months After Treatment Completion | Baseline: within 7 days before treatment start; Post-treatment: within 7 days after treatment completion; Follow-up assessments: at 1 month (±7 days), 2 months (±7 days), and 3 months (±7 days) after treatment completion.
  The number of suicide attempts will be assessed at five time points (baseline, post-treatment, and monthly during the 3-month follow-up) using the Columbia-Suicide Severity Rating Scale (C-SSRS), administered via in-person or telephone interview. Data will be cross-checked against available medical records as applicable.
Time to First Suicide Attempt After Treatment Completion | 1 month (±7 days), 2 months (±7 days), and 3 months (±7 days) after treatment completion.
  The number of days from treatment completion (end of Videoconference-Based Brief Cognitive Behavioral Therapy) to the first reported suicide attempt, assessed through monthly follow-up period (for example, using the Columbia-Suicide Severity Rating Scale, administered in person or by telephone).

SECONDARY OUTCOMES:
Intensity of suicidal ideation measured by Columbia-Suicide Severity Rating Scale (C-SSRS) | Baseline: ≤7 days before treatment start; Post-treatment: ≤7 days after treatment completion; Follow-up assessments: 1 month (±7 days), 2 months (±7 days), and 3 months (±7 days) after treatment completion.
  Suicidal ideation intensity will be assessed using the Intensity of Ideation items of the C-SSRS (frequency, duration, controllability, deterrents, and reasons for ideation), each scored from 0 to 5. Higher scores indicate greater ideation intensity.
Severity of suicidal ideation measured by Beck Scale for Suicide Ideation (SSI) | Baseline: ≤7 days before treatment start; Post-treatment: ≤7 days after treatment completion; Follow-up assessments: 1 month (±7 days), 2 months (±7 days), and 3 months (±7 days) after treatment completion.
  Suicidal ideation severity will be assessed using the Beck Scale for Suicide Ideation, a 19-item self-report questionnaire. Each item is scored from 0 to 2, producing a total score from 0 to 38. Higher scores indicate greater severity of suicidal ideation.
Change in depressive symptoms measured by Hamilton Depression Rating Scale (HAM-D-17) | Baseline: ≤7 days before treatment start; Post-treatment: ≤7 days after treatment completion; Follow-up assessments: 1 month (±7 days), 2 months (±7 days), and 3 months (±7 days) after treatment completion.
  Depressive symptom severity will be assessed at five time points using the 17-item Hamilton Depression Rating Scale. This clinician-administered semi-structured interview yields total scores ranging from 0 to 52, with higher scores indicating more severe depression.
Change in depressive symptoms measured by Beck Depression Inventory-II (BDI-II) | Baseline: ≤7 days before treatment start; Post-treatment: ≤7 days after treatment completion; Follow-up assessments: 1 month (±7 days), 2 months (±7 days), and 3 months (±7 days) after treatment completion.
  Depressive symptom severity will be assessed at five time points using the Beck Depression Inventory-II, a 21-item self-report questionnaire. Each item is scored from 0 to 3, yielding total scores from 0 to 63. Higher scores indicate greater symptom severity.
Change in hopelessness measured by the Beck Hopelessness Scale (BHS) | Baseline: ≤7 days before treatment start; Post-treatment: ≤7 days after treatment completion; Follow-up assessments: 1 month (±7 days), 2 months (±7 days), and 3 months (±7 days) after treatment completion.
  Change in the level of hopelessness will be assessed at five time points: baseline, post-treatment, and monthly for 3 months following treatment completion. Hopelessness will be measured using the Beck Hopelessness Scale (BHS), a 20-item self-report questionnaire designed to assess negative expectations about the future. Each item is scored dichotomously (True/False), with total scores ranging from 0 to 20. Higher scores indicate greater levels of hopelessness and have been associated with increased suicide risk.

OTHER OUTCOMES:
Consent rate (as an indicator of feasibility) | For each participant, from the time they are found eligible through screening until the time they provide informed consent and are randomized, during the study's active recruitment period (approximately 6 months).
  Consent rate will be used as a key feasibility indicator. It is defined as the percentage of eligible participants who provided informed consent and were randomized. The rate will be calculated by dividing the number of participants who consented and were randomized by the total number of eligible participants screened during the recruitment period.
Retention rate (as an indicator of feasibility) | From randomization: Baseline (≤7 days pre-start); Post-treatment (≤7 days post-completion); follow-ups at 1, 2, and 3 months (±7 days) after completion.
  Retention rate will be used as a key feasibility indicator. It is defined as the percentage of randomized participants who remained in the study and provided valid primary outcome data at each designated follow-up time point. The rate will be calculated by dividing the number of participants who completed the primary outcome assessment at each time point by the total number of participants randomized.
Adherence to treatment (as an indicator of feasibility) | From the first to the eighth scheduled treatment session, over the intervention period (approximately 4 weeks), for each participant assigned to the intervention group.
  Adherence to treatment will be used as a feasibility indicator. It is defined as the percentage of participants who attended all 8 scheduled treatment sessions. The rate will be calculated by dividing the number of participants who completed all sessions by the total number of participants assigned to the intervention group.
Death-Implicit Association Test (D-IAT) | Baseline: ≤7 days before treatment start; Post-treatment: ≤7 days after treatment completion; Follow-up assessments: 1 month (±7 days), 2 months (±7 days), and 3 months (±7 days) after treatment completion.
  Implicit identification with death will be assessed using the Death-Implicit Association Test (D-IAT), a computerized task measuring automatic associations between death-related concepts and the self. The Korean version of the D-IAT, validated for local use, consists of seven blocks administered via PsychoPy software. The outcome score (D-score) is computed using a standard scoring algorithm: a positive D-score indicates a stronger implicit association between death and self, while a negative score indicates a stronger association between life and self. Higher D-scores have been associated with increased risk of suicide attempts.
Anxiety symptoms measured by the Beck Anxiety Inventory (BAI) | Baseline: ≤7 days before treatment start; Post-treatment: ≤7 days after treatment completion; Follow-up assessments: 1 month (±7 days), 2 months (±7 days), and 3 months (±7 days) after treatment completion.
  Anxiety symptoms will be assessed at all scheduled time points using the Beck Anxiety Inventory (BAI), a 21-item self-report questionnaire. Each item is rated on a 0 to 3 scale, yielding a total score from 0 to 63. Higher scores indicate greater anxiety severity.
Emotion dysregulation measured by the Difficulties in Emotion Regulation Scale (DERS) | Baseline: ≤7 days before treatment start; Post-treatment: ≤7 days after treatment completion; Follow-up assessments: 1 month (±7 days), 2 months (±7 days), and 3 months (±7 days) after treatment completion.
  Emotion dysregulation will be assessed at all scheduled time points using the 35-item Korean version of the Difficulties in Emotion Regulation Scale (DERS). This self-report questionnaire measures six dimensions of emotion regulation difficulties: Nonacceptance of emotional responses, Difficulties engaging in goal-directed behavior, Impulse control difficulties, Lack of emotional awareness, Limited access to emotion regulation strategies, and Lack of emotional clarity. Each item is rated on a 5-point Likert scale from 1 to 5, with higher scores indicating greater difficulties in emotion regulation.
The Altman Self-Rating Mania Scale(ASRM) | Baseline: ≤7 days before treatment start; Post-treatment: ≤7 days after treatment completion; Follow-up assessments: 1 month (±7 days), 2 months (±7 days), and 3 months (±7 days) after treatment completion.
  Manic/hypomanic symptom severity will be assessed using the Altman Self-Rating Mania Scale (ASRM), a 5-item self-report questionnaire developed to measure the presence and severity of manic symptoms. Each item is rated from 0 to 4 based on symptom severity; higher scores indicate greater manic symptom severity.
Young Mania Rating Scale(YMRS) | Baseline: ≤7 days before treatment start; Post-treatment: ≤7 days after treatment completion; Follow-up assessments: 1 month (±7 days), 2 months (±7 days), and 3 months (±7 days) after treatment completion.
  Manic/hypomanic symptom severity will be assessed using the Young Mania Rating Scale (YMRS), an 11-item clinician-rated scale. Each item is rated on a 0-4 scale, with higher scores indicating greater manic symptom severity.
Distress tolerance measured by the Distress Intolerance Index | Baseline: ≤7 days before treatment start; Post-treatment: ≤7 days after treatment completion; Follow-up assessments: 1 month (±7 days), 2 months (±7 days), and 3 months (±7 days) after treatment completion.
  Distress tolerance will be assessed at all scheduled time points using the Distress Intolerance Index (DII), a 10-item self-report questionnaire. Each item is rated on a 5-point Likert scale from 0 (not at all like me) to 4 (very much like me), with total scores ranging from 0 to 40. Higher scores indicate lower distress tolerance.
Negative automatic thoughts measured by the Automatic Thoughts Questionnaire-Negative (ATQ-N) | Baseline: ≤7 days before treatment start; Post-treatment: ≤7 days after treatment completion; Follow-up assessments: 1 month (±7 days), 2 months (±7 days), and 3 months (±7 days) after treatment completion.
  Negative automatic thoughts will be assessed using the Automatic Thoughts Questionnaire-Negative (ATQ-N), a 30-item self-report measure. Participants rate how frequently they experienced each thought on a 5-point Likert scale from 1 (not at all) to 5 (all the time). Total scores range from 30 to 150, with higher scores indicating greater frequency of negative automatic thoughts.
Positive automatic thoughts measured by the Automatic Thoughts Questionnaire-Positive (ATQ-P) | Baseline: ≤7 days before treatment start; Post-treatment: ≤7 days after treatment completion; Follow-up assessments: 1 month (±7 days), 2 months (±7 days), and 3 months (±7 days) after treatment completion.
  Positive automatic thoughts will be assessed using the Automatic Thoughts Questionnaire-Positive (ATQ-P), a 30-item self-report measure. Each item is rated on a 5-point Likert scale from 1 (not at all) to 5 (all the time). Total scores range from 30 to 150, with higher scores indicating more frequent positive automatic thoughts.
Interpersonal needs measured by the Interpersonal Needs Questionnaire (INQ) | Baseline: ≤7 days before treatment start; Post-treatment: ≤7 days after treatment completion; Follow-up assessments: 1 month (±7 days), 2 months (±7 days), and 3 months (±7 days) after treatment completion.
  Interpersonal needs will be assessed using the Interpersonal Needs Questionnaire (INQ), a 15-item self-report measure designed to assess two constructs: perceived burdensomeness and thwarted belongingness. Each item is rated on a 7-point Likert scale from 1 (not at all true for me) to 7 (very true for me). Higher scores reflect greater interpersonal distress.
Fearlessness about death measured by the Acquired Capability for Suicide Scale - Fearlessness About Death (ACSS-FAD) | Baseline: ≤7 days before treatment start; Post-treatment: ≤7 days after treatment completion; Follow-up assessments: 1 month (±7 days), 2 months (±7 days), and 3 months (±7 days) after treatment completion.
  Fearlessness about death will be assessed using the Acquired Capability for Suicide Scale - Fearlessness About Death (ACSS-FAD), a 7-item self-report questionnaire. Each item is rated on a 5-point Likert scale from 0 (not at all like me) to 4 (very much like me), with higher scores indicating greater fearlessness about death.
Treatment satisfaction measured by the Client Satisfaction Questionnaire (CSQ-8) | Post-treatment (within 7 days after treatment completion), for participants in the intervention (V-BCBT) arm only.
  Treatment satisfaction will be assessed using the Client Satisfaction Questionnaire (CSQ-8), an 8-item self-report instrument rated on a 4-point Likert scale. The measure assesses satisfaction with treatment quality, perceived effectiveness, and willingness to reuse or recommend the intervention. Higher total scores indicate greater satisfaction.
Use and perceived helpfulness of intervention techniques measured by the Utility of Techniques (UT) questionnaire | Baseline: ≤7 days before treatment start; Post-treatment: ≤7 days after treatment completion; Follow-up assessments: 1 month (±7 days), 2 months (±7 days), and 3 months (±7 days) after treatment completion.
  The Utility of Techniques (UT) questionnaire will be used to assess participants' frequency of use and perceived helpfulness of specific intervention components. For each technique the participant reports having learned during the inpatient stay, they will rate frequency of use (from "not at all" to "more than 10 times per week") and helpfulness (if used, from "not at all" to "extremely"). Techniques include, for example, personalized safety planning tools and coping strategies taught during the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No